CLINICAL TRIAL: NCT05828641
Title: Comparison of Supination/Flexion Maneuver to Hyperpronation Maneuver in the Reduction of Radial Head Subluxations: A Randomized Clinical Trial
Brief Title: Comparison of Supination/Flexion Maneuver to Hyperpronation Maneuver
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: According to the results of the interim analysis when 50% of the targeted sample size was reached, a statistically significant benefit was detected with a large effect size in one treatment arm. For this reason, the study was terminated prematurely.
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan AKSEL, Associate Professor, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 211913807
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Emergencies; Orthopedics; Radial Head Subluxation
Keywords: Pediatric; pulled elbow; radial head subluxation; hyperpronation; supination-flexion; nursemaid's elbow; emergency medicine; supination flexion
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: This study is designed as parallel group randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The primary outcome accessors will be blinded to the study. They will not know which group is supination-flexion group or hyperpronation group from the data set. Group names will be included in the dataset as group 1 and group 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supination-flexion (Active Comparator): Supination-flexion maneuver will be applied in the treatment of patients in this group.
  Interventions: Procedure: Supination-flexion maneuver
- Hyperpronation (Active Comparator): Hyperpronation maneuver will be applied in the treatment of patients in this group.
  Interventions: Procedure: Hyperpronation maneuver

INTERVENTIONS:
Procedure: Supination-flexion maneuver — In the Supination-flexion group, the forearm will be supinated first, followed by full flexion of the elbow joint (Supination-flexion maneuver).
  Other Names: Supination flexion
  Arms: Supination-flexion
Procedure: Hyperpronation maneuver — In the hyperpronation group, the forearm will be pronated with the child's palm facing down (hyperpronation maneuver).
  Other Names: Hyper pronation
  Arms: Hyperpronation

SUMMARY:
This study is designed as a randomized controlled study. The investigators aim to compare the success of supination-flexion and hyperpronation maneuvers in the treatment of preschool children presenting to the emergency department with radial head subluxation.

All children aged 0-6 years, who are diagnosed with radial head subluxation secondary to traction of the forearm, had no evidence of direct trauma to the arm or fracture in the arm (no deformity, swelling, ecchymosis), had no history of musculoskeletal disease, and are approved to participate in the study by their legal guardians, will be included in the study. Patients who are considered to have radial head subluxation initially but had an X-ray performed by the physician and had a fracture in the arm will be excluded from the study.

In the study, patients will be randomized and assigned to two treatment groups: the supination-flexion group and the hyperpronation group. In the supination-flexion group, the forearm will be supinated first, followed by full flexion of the elbow joint. In the hyperpronation group, the forearm will be pronated with the child's palm facing down. In both groups, maneuvers will be performed by 3 emergency medicine specialists with at least 2 years of experience.

First-attempt failure is determined as the primary outcome of the study. Failure in the second attempt, ultimate failure, recurrence, patient satisfaction during the procedure, pain intensity (assessed by the Face, Legs, Activity, Cry, Consolability - FLACC pain scale), and treatment-related adverse events are determined as secondary outcomes of the study.

The investigators calculated the sample size and decided to include 117 patients in each group.

DETAILED DESCRIPTION:
INTRODUCTION Radial head subluxation also called nursemaid's elbow and pulled elbow, usually results from a sudden pull on the outstretched arm and is the most common cause of upper extremity injuries in preschool children. The diagnosis is made clinically and there is no need for routine imaging. The child complains of pain and refuses to use the affected arm. Radial head subluxation is treated with manual reduction of the subluxated radial head. Among the various reduction maneuvers available, the commonly used methods are supination-flexion and hyperpronation maneuvers.

The issue of which maneuver is more successful is still controversial. Supination-flexion is generally accepted as the standard maneuver and is the most preferred method. However, the hyperpronation technique was reported to be superior in a 2017 Cochrane review with 8 articles. But in a more recent randomized controlled trial on 152 patients it was reported that the supination-flexion maneuver was more successful. Controversial is not just the contradiction of previous study results. In addition, the quality of evidence is also controversial, as previous studies carry a high risk of bias. There is a serious risk of selection bias in most of the studies due to the lack or insufficiency of randomization or allocation concealment. Again, since there is no assessor blinding in the majority of the studies, the risk of detection bias is inevitable. Furthermore, in most of the previous randomized controlled trials, the sample size was not calculated. As a result, as highlighted in the Cochrane review, most previous randomized controlled trials, have a high risk of bias. The investigators think that well-planned, low-bias randomized controlled trials, are needed to answer this clinical question, both due to the high risk of bias in previous studies and conflicting results regarding which maneuver is superior in published reports.

In this randomized controlled study, the investigators aimed to compare the success of supination-flexion and hyperpronation maneuvers in the treatment of preschool children presenting to the emergency department with radial head subluxation.

METHODS This study will be conducted and reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) 2010 statement.

Design This parallel group open-label randomized controlled trial will be conducted between May 2023 and May 2024 in a tertiary education and research hospital.

Ethics committee approval was obtained from the local ethics committee of Umraniye Training and Research Hospital (Ethics Committee approval date: 21 March 2023, approval number: 211913807).

Population All children aged 0-6 years, who will be diagnosed with radial head subluxation secondary to traction of the forearm, had no evidence of direct trauma to the arm or fracture in the arm (no deformity, swelling, ecchymosis), had no history of musculoskeletal disease, and will be approved to participate in the study by their legal guardians, will be included in the study. Patients who are considered to have radial head subluxation initially but had an X-ray performed by the physician and had a fracture in the arm will be excluded from the study.

Diagnosis The patients will be diagnosed with radial head subluxation clinically, and if the child shows symptoms of pain after traction on the arm and refuses to use the arm on that side, the diagnosis of radial head subluxation will be made. In cases where routine imaging will not be requested, but the history and physical examination are not clear, imaging will be requested at the discretion of the physician managing the patient.

Interventions In the study, patients will be randomized and assigned to two treatment groups: the supination-flexion group and the hyperpronation group. In the supination-flexion group, the forearm will be supinated first, followed by full flexion of the elbow joint. In the hyperpronation group, the forearm will be pronated with the child's palm facing down. In both groups, maneuvers will be performed by 3 emergency medicine specialists with at least 2 years of experience.

Outcome measurements First-attempt failure is determined as the primary outcome of the study. 10 minutes after the procedure, the patient will be re-examined and the success of the treatment will be evaluated. If additional treatment is needed or if the child still avoids using his/her arm after the procedure, it will be considered a treatment failure. If the participant's pain decreases and the participant can use the effected arm easily, the maneuver will be considered successful.

Failure in the second attempt, ultimate failure (failure after the third reduction attempt), recurrence (re-admission with radial head subluxation in the same arm within 72 hours), and pain intensity of the patient (will be assessed by the Face, Legs, Activity, Cry, Consolability pain scale (FLACC)), treatment-related adverse events (fracture of the forearm, hyperemia, vascular injury, nerve injury after the first attempt) are determined as secondary outcomes of the study.

Randomization Randomization will be done via www.randomizer.org and in 6 blocks. Treatment allocation will be concealed and performed by means of a computerized balanced allocation method.

Blinding The study is not suitable for blindness since two different maneuvers will be applied as intervention and therefore it was designed as open-label. However, the accessors will be blinded to the study.

Sample Size Calculation G*Power 3.1.9.6 software was used for sample size calculation. In studies comparing two reduction methods in the literature, the failure rate at the first attempt was reported as 16.2-34.2% in the supination-flexion group and 4.4-20.9% in the hyperpronation group. In addition, in the Cochrane review, which compared both reduction methods and was published in 2017, the failure rate in the supination-flexion group was reported as 26.4%. The supination-flexion group was considered the control group, and a 15% reduction in failure was considered clinically significant. To detect such a difference, it was calculated that 106 patients should be included in each group using a two-sided alpha value of 5% and a power of 80%. Finally, considering the potential data loss of 10%, it is decided to include 117 patients in each group.

Statistical analysis SPSS 26 (IBM Corp. Released 2019. IBM SPSS Statistics for Windows, Version 26.0. Armonk, NY: IBM Corp.) will be used for statistical analysis. The normal distribution of continuous data will be determined by the Shapiro-Wilk test and histograms. Normally distributed data will be expressed as mean and standard deviation and non-normally distributed data will be expressed as median and quartiles. The Student-T test will be used for the comparison between groups for continuous data with normal distribution, and the Mann-Whitney U test for those without normal distribution. Categorical data, such as primary outcome treatment failure rates, will be expressed as frequency and percentage, and the Chi-square test will be used for group comparison for categorical variables (Fisher's exact test where necessary).

A statistically significant level of p<0.05 was accepted.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of radial head subluxation
* No evidence of direct trauma to the arm
* No fracture in the arm
* No history of musculoskeletal disease

Exclusion Criteria:

-Refusing to participate in the study

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Rate of first attempt failure | 10 minutes after the first-attempt, the outcome will be evaluated.
  After the first attempt (the maneuver according to group), the patient will re-examined and the success of the treatment will be evaluated. If additional treatment was needed or if the child still avoided using his/her arm after the procedure, it was considered as treatment failure

SECONDARY OUTCOMES:
Rate of second attempt failure | 10 minutes after the second-attempt, the outcome will be evaluated.
  After the second attempt (same maneuver as the first maneuver), the patient will re-examined and the success of the treatment will be evaluated. If additional treatment was needed or if the child still avoided using his/her arm after the procedure, it was considered as treatment failure
Rate of third attempt failure (ultimate failure) | 10 minutes after the third-attempt, the outcome will be evaluated.
  In the presence of treatment failure despite performing the same maneuver 3 times, this will be considered as ultimate failure.
Number of patients presenting with recurrence of radial head subluxation | 72 hours after of first admission with same diagnosis.
  Re-admission with radial head subluxation in the same arm within 72 hours.
Pain intensity of the patients during the first attempt of the maneuver | Just before (1 minute) and during the first attempt of the maneuver.
  The pain intensity of the patient will be assessed by the Face, Legs, Activity, Cry, Consolability pain scale (FLACC). Higher scores mean worse outcome.
  Assessment of the score:
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Adverse events detected during the first attempt of the maneuver | Side effect assessment will begin immediately after the reduction maneuver is performed. The patient will be followed up for side effects for a week and any side effects seen during this period will be recorded.
  Fracture of the forearm, hyperemia, vascular injury, nerve injury after the first attempt.

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choung W, Heinrich SD. Acute annular ligament interposition into the radiocapitellar joint in children (nursemaid's elbow). J Pediatr Orthop. 1995 Jul-Aug;15(4):454-6. doi: 10.1097/01241398-199507000-00008. PMID 7560033
- [Background] Hanes L, McLaughlin R, Ornstein AE. Suspected Radial Head Subluxation in Infants: The Need for Radiologic Evaluation. Pediatr Emerg Care. 2021 Jan 1;37(1):e58-e59. doi: 10.1097/PEC.0000000000001848. PMID 31283721
- [Background] Krul M, van der Wouden JC, Kruithof EJ, van Suijlekom-Smit LW, Koes BW. Manipulative interventions for reducing pulled elbow in young children. Cochrane Database Syst Rev. 2017 Jul 28;7(7):CD007759. doi: 10.1002/14651858.CD007759.pub4. PMID 28753234
- [Background] Porozan S, Forouzan A, Hassanzadeh R. Hyperpronation versus Supination-Flexion in Radial Head Subluxation Reduction: A Randomized Controlled Trial. J Pediatr Intensive Care. 2020 Dec;9(4):256-260. doi: 10.1055/s-0040-1709703. Epub 2020 Apr 29. PMID 33133740
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Gunaydin YK, Katirci Y, Duymaz H, Vural K, Halhalli HC, Akcil M, Coskun F. Comparison of success and pain levels of supination-flexion and hyperpronation maneuvers in childhood nursemaid's elbow cases. Am J Emerg Med. 2013 Jul;31(7):1078-81. doi: 10.1016/j.ajem.2013.04.006. Epub 2013 May 20. PMID 23702058
- [Background] McDonald J, Whitelaw C, Goldsmith LJ. Radial head subluxation: comparing two methods of reduction. Acad Emerg Med. 1999 Jul;6(7):715-8. doi: 10.1111/j.1553-2712.1999.tb00440.x. PMID 10433531
- [Background] Green DA, Linares MY, Garcia Pena BM, Greenberg B, Baker RL. Randomized comparison of pain perception during radial head subluxation reduction using supination-flexion or forced pronation. Pediatr Emerg Care. 2006 Apr;22(4):235-8. doi: 10.1097/01.pec.0000210172.17892.a1. PMID 16651912
- [Background] Guzel M, Salt O, Demir MT, Akdemir HU, Durukan P, Yalcin A. Comparison of hyperpronation and supination-flexion techniques in children presented to emergency department with painful pronation. Niger J Clin Pract. 2014 Mar-Apr;17(2):201-4. doi: 10.4103/1119-3077.127557. PMID 24553032
- [Derived] Aksel G, Kuka B, Islam MM, Demirkapi F, Ozturk I, Islek OM, Ademoglu E, Eroglu SE, Satici MO, Ozdemir S. Comparison of supination/flexion maneuver to hyperpronation maneuver in the reduction of radial head subluxations: A randomized clinical trial. Am J Emerg Med. 2025 Feb;88:29-33. doi: 10.1016/j.ajem.2024.11.026. Epub 2024 Nov 18. PMID 39579408